CLINICAL TRIAL: NCT02157545
Title: The Dose-response Relationship of Rocuronium in Patients Taking Pyridostigmine Preoperatively Compared With Age and Sex Matched Controls
Brief Title: The Dose-Response Relationship of Rocuronium in Patients Taking Pyridostigmine
Status: Withdrawn | Type: Observational
Why Stopped: No eligible subjects identified. Study closed with IRB.
Sponsor: Shashi Bhatt, MD (Other)
Responsible Party: Sponsor-Investigator, Shashi Bhatt, MD, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Other Study IDs: Pyridostigmine
Record Dates: First submitted 2014-05-21; First posted 2014-06-06 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Muscle Relaxants
Keywords: muscle relaxants; pyridostigmine; pharmacodynamics; potency
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pyridostigmine: administration of rocuronium to determine its potency.
- control arm (no pyridostigmine): determination of potency of rocuronium in patients not taking pyridostigmine

SUMMARY:
Pyridostigmine is a medication that is used in certain heart rate and blood pressure conditions. This medication, as a side effect, is known to also cause changes in the junction between a nerve and muscle. The changes caused at the nerve muscle junction by pyridostigmine could alter the effect of muscle relaxants (a medication used during surgery and anesthesia). The investigators are conducting this study to see whether patients taking pyridostigmine are more or less sensitive to rocuronium (a muscle relaxing medication used during surgery).

DETAILED DESCRIPTION:
No subjects enrolled. No data collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who take pyridostigmine for any reason or those who are matched by age, sex and weight to subjects taking pyridostigmine
* Patients who will be administered rocuronium during elective procedures as standard clinical care.

Exclusion Criteria:

* Allergy to rocuronium
* Known neuromuscular disorder, patients suffering from myasthenia gravis
* Subjects taking medications known to impact neuromuscular transmission (ex. gentamicin).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects taking pyridostigmine for any reason who are scheduled for surgery under general anesthia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Dose of the muscle relaxant rocuronium that will lead to 50% decrease in the force of the evoked muscle contraction in patients taking pyridostigmine. | 12 months
  Rocuronium used to produce muscle weakness or paralysis during surgery. Its potency is measured as ED50, the dose necessary to cause a 50% reduction in the force of evoked muscle contraction. We intend to determine this measure of potency (ED50 for rocuronium) in patients taking pyridostigmine and compare it with control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Shashi Bhatt, MD, Principal Investigator — University of Toledo Health Science Campus
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data collected.